CLINICAL TRIAL: NCT00372398
Title: Premature Coronary Atherosclerosis in Scleroderma: A Case Control Study
Brief Title: Premature Coronary Atherosclerosis in Scleroderma
Status: Completed | Type: Observational
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: CC Mok, Tuen Mun Hospital, Hong Kong
Other Study IDs: NTWC/CREC/429/06
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Scleroderma
Keywords: scleroderma; sclerosis; atherosclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Sclerosis; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this trial is to study the proportion of scleroderma patients who suffer from asymptomatic coronary atherosclerosis compared to healthy controls.

DETAILED DESCRIPTION:
Coronary calcium scores will be obtained from a group of patients with scleroderma and a group of controls. Comparison of the calcium scores will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Fulfillment of the American College of Rheumatology (ACR) criteria for the classification of scleroderma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: scleroderma patients
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD FRCP, Principal Investigator — Tuen Mun Hospital Hong Kong
Locations (1):
- Tuen Mun Hospital, Hong Kong, Hong Kong